CLINICAL TRIAL: NCT05842187
Title: A Multi-center, Prospective, Exploratory Study Evaluating the Effectiveness of Treatment Regimens for Metastatic Pancreatic and Gastric Cancer Guided by in Vitro Drug Sensitivity Testing of Tumor Organoids
Brief Title: In Vitro Organoid Drug Sensitivity-Guided Treatment for Metastatic Pancreatic and Gastric Cancer
Acronym: ODYSSEY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianzhen Shan, MD (Other)
Responsible Party: Sponsor-Investigator, Jianzhen Shan, MD, Director of Medical Oncology Department (4), First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20230001C-R1
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Cancer; Gastric Cancer
Keywords: pancreatic cancer; gastric cancer; organoid; drug sensitivity
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organoid generation (Experimental): All patients will be included in a single-arm. Participants will undergo biopsy of tumor tissue for subsequent organoid generation
  Interventions: Procedure: Biopsy of tumor tissue for organoid culture

INTERVENTIONS:
Procedure: Biopsy of tumor tissue for organoid culture — By collecting fresh tumor tissues (including ascites, pleural effusion, biopsy tissues, palliative surgery specimens, etc.) and culturing them into organoids in vitro, this study conducts drug sensitivity tests on various clinically approved drugs. The most sensitive drug for the patient is selected for treatment, and the study aims to evaluate the clinical effectiveness of the drug and its consistency with in vitro organoid drug sensitivity.

SUMMARY:
The goal of this study is to evaluate the consistency between in vitro tumor organoid drug sensitivity and the therapeutic efficacy of in vivo drug treatment.

Participants are required to provide one of fresh tumor tissues (including ascites, pleural effusion, biopsy tissues, palliative surgery specimens, etc.) for the purpose of culturing tumor organoids.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years old.
2. Metastatic pancreatic cancer with progression after second-line or higher treatment, metastatic gastric cancer with progression after third-line or higher treatment, or metastatic pancreatic or gastric cancer patients who cannot tolerate standard treatment regimens.
3. Able to provide fresh tumor tissue specimens for organoid culture, including: ascites, pleural effusion, tumor biopsy tissues, tumor surgical specimens, etc.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2.
5. Adequate organ function, including the following:

   * Bone marrow: Absolute neutrophil count (ANC) in peripheral blood ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, hemoglobin ≥ 80 g/L.
   * Liver: Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) ≤ 3 times ULN. If liver metastases are present, aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) ≤ 5 times ULN.
   * Kidney: Creatinine clearance ≥ 45 mL/min (using the standard Cockcroft-Gault formula) or ≤ 1.5 times ULN.
6. At least one measurable or evaluable lesion.
7. For women: Must be sterilized, postmenopausal, or using highly effective contraception during treatment and for 3 months after treatment; must not be pregnant or breastfeeding during treatment.
8. Patient compliance and geographic proximity to ensure adequate follow-up.

Exclusion Criteria:

1. Any unstable systemic disease (including systemic active infections requiring treatment, liver disease, kidney disease, or metabolic diseases, acute cerebral infarction or cerebral hemorrhage, etc.) that, in the investigator's judgment, may impair patient safety or the patient's ability to complete the study due to severe comorbidities.
2. Significant cardiovascular events: Congestive heart failure > NYHA class 2; unstable angina, active coronary artery disease (CAD) (myocardial infarction more than 1 year before the study is allowed); severe arrhythmias requiring treatment (use of beta-blockers or digoxin is allowed) or uncontrolled hypertension, etc.
3. Significant history of neurological or psychiatric disorders, including epilepsy, dementia, etc.
4. Pregnant or breastfeeding women; those of childbearing potential who are unwilling or unable to use effective contraception.
5. Other situations that the investigator judges may affect the conduct and determination of the clinical research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS (Progressive free survival) | 6 months
  The time from initiation of treatment to the occurrence of disease progression or death.

SECONDARY OUTCOMES:
DCR (Disease control rate) | 6 months
  The percentage of patients who have achieved complete response, partial response and stable disease to a therapeutic intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No